CLINICAL TRIAL: NCT04095260
Title: Identification of Neuromusculoskeletal Variables Associated With Injury Risk and Performance in High School Athletes.
Status: Not yet recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0135
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high school athletes: High school athletes, ages 14 to 18, who are participating in an organized sports training program.
  Interventions: Other: Pre-season strength and conditioning program

INTERVENTIONS:
Other: Pre-season strength and conditioning program — The structured physical performance assessment will include functional movement testing, motor coordination testing, joint mobility screen, muscle strength testing, and agility performance testing. These measures will assess the effectiveness of pre-season strength and conditioning program to reduce musculoskeletal impairments and increase resistance to injury.
  Other Names: pre and post physical performance testing following a high school based strength and conditioning training program

SUMMARY:
The purpose of this study is to complete a neuromuscular performance assessment of high school athletes who are participating in school based pre-season strength and performance training program. The performance assessment will screen for existing muscle imbalances and strength deficits known to increase risk for sports injury, and provide a baseline performance measurement. Athletes will be measured before the start of the program and then again at the end of the pre-season training period to measure changes in motor coordination, muscle strength, and performance and injury risk category. Internal and external training load will be measured weekly during the training program to track intensity of the training program. In addition to the pre and post measurements, sports injury occurrence and time away from sports participation will be tracked throughout the sport season/school year to evaluate training program outcomes and accuracy of risk assessment.

DETAILED DESCRIPTION:
This study involves a test - re-test design. Subjects will be tested in their physical performance. These measures include a general assessment of joint mobility, muscle strength, motor coordination, and performance assessment utilizing functional movement screens. The physical examination is similar to a physical examination performed clinically in sports performance testing and also in the practice of Physical Therapy. The initial baseline measure will provide objective scores that can be utilized to assess for change over time. Additional information to be gathered includes demographic information on the subject including age, previous injury history, and level of exposure to physical performance training. These variables are associated with injury risk and also impact the potential for change with physical performance training. In addition, information on mental factors including stress, fear of failure, and burnout will be collected. It is hypothesized that these variables also factor into athletic performance. It is not known how these variables impact injury risk. Information on training load will be gathered weekly during the training period. Training load has a direct impact on muscle performance, and is hypothesized to impact injury risk. The subjects will be re-tested at the end of the training period to measure changes in physical performance and injury risk.

Project Procedures

Study population: High school athletes, ages 14 to 18, who are participating in an organized sports training program. The target subject enrollment is 250 high school athletes.

Inclusion criteria will be athletes who have completed a pre-participation sports physical, are enrolled in a sports elective or a member of a sports team, and have volunteered to participate in the study providing both verbal and written consent.

Exclusion criteria for participation include athletes who have not submitted a pre-participation sports physical to the high school training staff, student athletes who are currently suffering from an acute neuromusculoskeletal injury with restrictions on athletic participation, an athlete who has undergone surgery within a 3 month period of the program start date, an athlete who presents with a cardiovascular condition that would exclude exercise participation (systolic BP > 180, diastolic BP > 100), or athletes who are currently pregnant.

Study Methodology

Participants will complete a self-report questionnaire collecting demographic data including age, gender, primary and secondary sport activity, and previous injury history. Participants will also complete the Perceived Stress Scale to measure self-appraised stress, the Sports Mental Training Questionnaire to measure mental preparation skills, and the Athlete Burnout Questionnaire to assess emotional/physical exhaustion at the beginning and end of the 8 week program to assess psychological stressors associated with sport participation that may impact motivation to participate and perceived internal training load.

The structured physical performance assessment will include functional movement testing, motor coordination testing, joint mobility screen, muscle strength testing, and agility performance testing. Video analysis will be included with the functional movement testing utilizing software to assess reliability of the neuromuscular impairment screen.

Research project specific measures:

Functional movement testing includes:

1. Forward flexion/hinge
2. Standing trunk rotation
3. Bilateral squat
4. Forward lunge
5. Lateral lunge
6. Lower extremity functional reach test
7. Upper extremity movement pattern (shoulder mobility test)
8. Quadruped trunk rotary stability test

Mobility testing includes:

1. Ankle mobility testing (DF, PF, IV, EV, first ray extension)
2. Hip mobility testing (flexion, extension, abduction, IR, ER)
3. Cervical mobility testing (flexion, extension, side bending, rotation, flexion rotation
4. Thoracic mobility testing (seated trunk rotation)
5. Shoulder mobility testing (flexion with scapular mobility assessment, abduction with scapular mobility assessment, IR, ER)
6. Elbow mobility testing (flexion, extension, supination, pronation)
7. Wrist mobility (flexion, extension)

Muscle strength testing:

1. Hip strength (flexion, extension, abduction, ER, IR)
2. Knee strength (flexion, extension)
3. Ankle strength (PF, IV, EV)
4. Shoulder strength (IR, ER, AB)
5. Scapular strength (middle trap, lower trap)
6. Elbow strength (flexion, extension)

Performance testing:

1. Jump testing (bilateral long jump, unilateral jump, drop box jump)
2. Upper extremity closed chain reach testing
3. Shuttle run

Intrinsic and Extrinsic training load will be recorded weekly for subjects participating in the research study. Data will be utilized to calculate the training load associated with the school based strength and conditioning training program.

ELIGIBILITY:
Inclusion Criteria:

* athletes who have completed a pre-participation sports physical
* are enrolled in a sports elective or a member of a sports team
* have volunteered to participate in the study providing both verbal and written consent.

Exclusion Criteria:

* athletes who have not submitted a pre-participation sports physical to the high school training staff
* student athletes who are currently suffering from an acute neuromusculoskeletal injury with restrictions on athletic participation
* an athlete who has undergone surgery within a 3 month period of the program start date
* an athlete who presents with a cardiovascular condition that would exclude exercise participation (systolic BP > 180, diastolic BP > 100)
* an athletes who are currently pregnant.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: High school athletes, ages 14 to 18, who are participating in an organized sports training program. The target subject enrollment is 250 high school athletes.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2028-08-01 (Estimated); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in baseline movement quality as measured by the Selective Functional Movement Assessment (SFMA). | Pre (initial baseline), and after week 8 of preseason strength and condition training program
  The Selective Functional Movement Assessment is an assessment to score movement quality on 7 functional movements. The movement is categorically scored as: Functional and not painful (FN); Functional and painful (FP); Dysfunctional and not painful (DN); Dysfunctional and painful (DP)
Change in muscle strength testing as measured by hand held dynamometer. | Pre (initial baseline) and after week 8 of preseason strength and condition training program
  Hand held dynamometer measures isometric force production in kilograms or pounds.
Change in baseline movement quality as measured by the Anterior reach of the Y Balance Test. | Pre (initial baseline) and after week 8 of preseason strength and condition training program
  The Anterior reach of the Y Balance Test measures distance of limb reach in centimeters. Distance is compared from one side to the other to assess for symmetry. A difference of > 4cm is a positive risk factor for lower extremity injury.
Change in baseline in motor performance as measured by the Single Leg Hop jump distance. | Pre (initial baseline) and after week 8 of preseason strength and condition training program
  Single leg hop test measures hop distance in centimeters. Distance hopped is compared between limbs, comparing strength and power symmetry between the two limbs.
Change in baseline in motor performance as measured by the Modified T-Test drill completion time (seconds). | Pre (initial baseline) and after week 8 of preseason strength and condition training program
  The Modified T-Test is an agility test that incorporates quick direction changes in a defined pattern. The test is measured in seconds. A reduction in the time to complete the drill represents improved motor performance and power.

SECONDARY OUTCOMES:
Number of participants who experience a musculoskeletal sports related injury. | End of study (1 year)
  Measuring occurrence of musculoskeletal injury that is reported by the athlete and/or impacts participation practice or playing time during the training and competition season. Number of missed days of practice and or sports competition will be recorded.
Intrinsic training load as measured by perceived effort of the training session (Rate of Perceived Exertion Scale) | Weekly, for 8 weeks during the strength and conditioning training program
  Rate of Perceived Exertion Scale is a 0 to 10 scale that measures the perceived difficulty of a training sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Janna M McGaugh, ScD, Principal Investigator — UTMB
Locations (1):
- Clear Falls High School, League City, Texas, United States

IPD SHARING:
Plan to Share IPD: No